CLINICAL TRIAL: NCT06694701
Title: Emapalumab Treatment For Anticipated Clinical Benefit In Sepsis Driven By The Interferon-Gamma Endotype (The EMBRACE Trial)
Acronym: EMBRACE
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hellenic Institute for the Study of Sepsis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EMBRACE; 2024-515255-38-00 (EU CTIS Number)
Record Dates: First submitted 2024-11-13; First posted 2024-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-03

CONDITIONS: Sepsis
Keywords: Severe infections; IFNγ; IFNγ-Drive Sepsis; emapalumab; interferon-gamma
MeSH Terms: conditions — Sepsis; Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Placebo (Placebo Comparator): Standard-of-care (SoC) treatment and placebo drug.
  Interventions: Drug: Placebo
- Emapalumab Group 1 (Active Comparator): SoC treatment and a low dose of emapalumab.
  Interventions: Drug: Emapalumab-Izsg
- Emapalumab Group 2 (Active Comparator): SoC treatment and a high dose of emapalumab.
  Interventions: Drug: Emapalumab-Izsg

INTERVENTIONS:
Drug: Emapalumab-Izsg — The drug is administered at a dose of 6mg/kg of body weight on day 0 and repeated dosing of 3mg/kg of body weight is provisioned for days 3, 6, 9, 12, 15, 19, 23 and 27 provided that the stopping rule does not apply.
  Other Names: Emapalumab Group 1
  Arms: Emapalumab Group 1
Drug: Emapalumab-Izsg — The drug is administered at a dose of 6mg/kg of body weight on day 0, 6mg/kg of body weight on day 3, 6mg/kg of body weight on day 6 and repeated dosing of 3mg/kg of body weight is provisioned for days 9, 12, 15, 19, 23 and 27 provided that the stopping rule does not apply.
  Other Names: Emapalumab Group 2
  Arms: Emapalumab Group 2
Drug: Placebo — 250ml of 0.9% sodium chloride. The drug is administered on day 0 and repeated dosing is provisioned for days 3, 6, 9, 12, 15, 19, 23 and 27 provided that the stopping rule does not apply
  Arms: Placebo

SUMMARY:
EMBRACE is a double-blind, randomized, placebo-controlled, phase IIa study that will be conducted in multiple Intensive Care Units (ICUs) and departments of Internal Medicine across Greece. It aims to investigate if treatment with emapalumab, a monoclonal antibody which blocks IFNγ, may improve the outcome of patients with sepsis driven by the IDS (endotype of IFNγ-driven sepsis) endotype. EMBRACE also aims to identify the best dosing regimen of emapalumab for the management of IDS.

DETAILED DESCRIPTION:
The EMBRACE trial aims to generate proof-of-concept if treatment with emapalumab, a monoclonal antibody which blocks IFNγ signaling, may improve the outcome of patients with sepsis driven by the IDS endotype. In EMBRACE, two different dose regimens of emapalumab are administered in order to: a) investigate which dose regimen may provide most of efficacy in the decrease of SOFA score, a new endpoint for sepsis suggested already by others; b) investigate which dose regimen better attains the pharmacodynamic goal of emapalumab defined as the decrease of blood CXCL9; and c) compare the efficacy of the two dose regimens with placebo treated patients.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent
* Adults (≥18 years) of male or female sex
* Diagnosis of community-acquired pneumonia (CAP), hospital-acquired pneumonia (HAP), ventilator-associated pneumonia (VAP), intrabdominal infection (IAI), acute pyelonephritis (AP), primary bloodstream infection (BSI) and viral respiratory infections.
* Sepsis defined by the Sepsis-3 definitions. This is defined as any new infection which is accompanied by an increase of the total baseline SOFA score by at least 2 points. The total baseline SOFA score is calculated by the medical comorbidities and by the evaluation of clinical variables before the sepsis episode in the case of hospital-acquired sepsis. In the case of patients with unknown baseline SOFA score, sepsis is defined as any new infection accompanied by total SOFA score 2 or more.
* Willingness to use effective contraceptive methods during the period from the start of the study drug to 6 months after the administration of the last dose of the study drug, in patients of reproductive age.
* Serological documentation of IDS defined as detectable blood IFNγ and CXCL9 more than 2,200 pg/ml. IFNγ and CXCL9 are measured in the central study lab by an enzyme immunosorbent assay.
* Absence of sepsis-induced immunoparalysis (SII). This is defined as ≥8000 of HLA-DR receptors on CD45/CD14-monocytes measured by flow-cytometry in the central lab using the BD™ fluorescence assay9.

Exclusion Criteria:

* Body weight more than 104 kg
* Intake of any other biological during the last 30 days prior screening except for the intake of anakinra or tocilizumab for patients with active infection by SARS-CoV-2
* Intake of any Janus kinase inhibitors during the last 30 days prior screening except for the intake of baricitinib for patients with active infection by SARS-CoV-2
* Known active infection by Mycobacterium tuberculosis or other mycobacteria. These patients may be enrolled in the trial if treatment against infection by Mycobacterium tuberculosis or other mycobacteria has been initiated
* Known active infection by VZV (varicella zoster virus) or by Histoplasma capsulatum or by Leishmania spp. These patients may be enrolled in the trial if treatment against infection by VZV or Histoplasma capsulatum has been initiated
* Known active infection by the hepatitis B virus, by the hepatitis C virus and by cytomegalovirus
* Vaccination the last 12 weeks before screening with BCG vaccine
* Vaccination with any live or attenuated live vaccine (other than BCG) the last 12 weeks before screening
* Known allergy or hypersensitivity reactions to emapalumab
* Patients living with the human immunodeficiency virus (HIV)
* Patients with stage IV solid or hematologic malignancy
* Patients with neutropenia (less than 1,000 neutrophils/mm3)
* Patients transplanted for solid organ or stem cells
* Pregnancy or lactation
* Participation in any other interventional trial the last 28 days prior to day 1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-03-22 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Decrease of SOFA score by the end-of-treatment | From enrollment to the end of treatment of the study drug for each of the study participants, ranging from 2 to 29 days.
  The study primary endpoint is the decrease of SOFA score by the end-of-treatment (EOT). This is defined as either a) at least 1.4 points decrease of mean SOFA score calculated between days 1 and EOT from SOFA score of day 0; OR b) at least 2 points decrease of SOFA at EOT from day 0.

SECONDARY OUTCOMES:
The rate of serious TEAEs and non-serious TEAEs | From enrollment to the end of observation of each of the study participants, which is 120 days plus or minus 3 days, after each participant's enrollment.
  Comparison of the rate of serious TEAEs and non-serious TEAEs between the three groups of treatment.
The number of doses required in each group to achieve the SOFA score response by the EOT. | From enrollment to the end of treatment of the study drug for each of the study participants, ranging from 2 to 29 days.
The change of the SOFA score from day 0 until day 7 | From enrollment (day 0) to 8 days after enrollment (day 7).
  Comparison of the change of the SOFA score from day 0 until day 7
28-day mortality | From enrollment to 28 days after enrollment.
The change of the SOFA score from 0 until day 28 | From enrollment to 28 days after enrollment.
  Comparison of the change of the SOFA score from 0 until day 28
The change of the SOFA score from 0 until EOT | From enrollment to the end of treatment of the study drug for each of the study participants, ranging from 2 to 29 days.
  Comparison of the change of the SOFA score from 0 until EOT
The pharmacokinetics of emapalumab | From enrollment to the end of treatment of the study drug for each of the study participants, ranging from 2 to 29 days.
  Comparison of the pharmacokinetics of emapalumab
The need to stop the study drug due to drop of the number of HLA-DR receptors on CD14-monocytes. | From enrollment to the end of treatment of the study drug for each of the study participants, ranging from 2 to 29 days.
  Comparison of the need to stop the study drug due to drop of the number of HLA-DR receptors on CD14-monocytes.
The circulating concentrations of IL-6, ferritin, IFNγ and CXCL9 over the days of treatment | From enrollment to the end of treatment of the study drug for each of the study participants, ranging from 2 to 29 days.
  Comparison of the circulating concentrations of IL-6, ferritin, IFNγ and CXCL9 over the days of treatment

OTHER OUTCOMES:
Comparison between the three groups of treatment for the proteomic profile over treatment | From enrollment to the end of treatment of the study drug for each of the study participants, ranging from 2 to 29 days.
The comparisons between the three groups of treatment for the change of the transcriptomic profile over treatment | From enrollment to the end of treatment of the study drug for each of the study participants, ranging from 2 to 29 days.
The diagnostic performance of the point-of-care SepsisLoop for SII compared to the absolute count of HLA-DR receptor on CD45/CD14-monocytes. | From enrollment to the end of treatment of the study drug for each of the study participants, ranging from 2 to 29 days.
The clinical data and bedside biomarker levels at screening for the potential development of a diagnostic tool classifying the study population into IDS | From enrollment to the end of treatment of the study drug for each of the study participants, ranging from 2 to 29 days.
The prognostic biomarker levels at screening classifying the Sepsis population in different subgroups | From enrollment to the end of treatment of the study drug for each of the study participants, ranging from 2 to 29 days.

CONTACTS AND LOCATIONS:
Overall Officials: Evangelos Giamarellos-Bourboulis, Study Chair — Hellenic Institute for the Studies of Sepsis
Locations (24):
- Greece (24):
  - 1st Department of Internal Medicine, Thriasio Elefsis General Hospital, Elefsina, Attica
  - Clinic of Intensive Care and Pulmonary Diseases, Aghioi Anargyroi Kifissia General Oncologic Hospital, Kifissia, Attica
  - Intensive Care Unit, University General Hospital of Heraklion, Heraklion, Crete
  - Intensive Care Unit, Alexandroupolis University General Hospital, Alexandroupoli
  - 3rd University Department of Internal Medicine, Sotiria Chest Diseases Athens General Hospital, Athens
  - 4th Department of Internal Medicine, ATTIKON University General Hospital, Athens
  - Intensive Care Unit I, KAT Attica General Hospital, Athens
  - Intensive Care Unit of 1st University Department Respiratory Medicine, Sotiria Chest Diseases Athens General Hospital, Athens
  - Intensive Care Unit of Center for Respiratory Failure, Sotiria Chest Diseases Athens General Hospital, Athens
  - Intensive Care Unit, Asklipieio Voulas General Hospital, Athens
  - Intensive Care Unit, Ippokrateio Athens General Hospital, Athens
  - Intensive Care Unit, Korgialeneio-Benakeio HRC Athens General Hospital, Athens
  - Intensive Care Unit, Laiko Athens General Hospital, Athens
  - New Multivalent Intensive Care Unit, Sotiria Chest Diseases Athens General Hospital, Athens
  - Ηigh Dependency Unit of Department of Clinical Therapeutics, Alexandra Athens General Hospital, Athens
  - Intensive Care Unit, Patras University General Hospital, Pátrai
  - 1st Intensive Care Unit, G. Papanikolaou Thessaloniki General Hospital, Thessaloniki
  - Department of Anesthesiology and Intensive Care, AHEPA Thessaloniki University General Hospital, Thessaloniki
  - Intensive Care Unit, 424 General Military Training Hospital, Thessaloniki
  - Intensive Care Unit, Aghios Dimitrios Thessaloniki General Hospital, Thessaloniki
  - Intensive Care Unit, G. Gennimatas Thessaloniki General Hospital, Thessaloniki
  - Intensive Care Unit, Ippokrateio Thessaloniki General Hospital, Thessaloniki
  - Intensive Care Unit, Papageorgiou Thessaloniki General Hospital, Thessaloniki
  - Intensive Care Unit, Theageneio Thessaloniki Cancer Hospital, Thessaloniki